CLINICAL TRIAL: NCT01922687
Title: Amlodipine Plus/Minus Atorvastatin for Protection of Arteries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Institute of Hypertension (Other)
Responsible Party: Principal Investigator, Yan Yang, Attending physician, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruijin2010No.14
Record Dates: First submitted 2013-07-30; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Arterial and Arteriolar Disorders
MeSH Terms: interventions — Amlodipine; Atorvastatin; amlodipine, atorvastatin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amlodipine Plus Atorvastatin (Caduet) (Experimental): amlodipine plus atorvastatin in a single tablet (Caduet, Pfizer, USA) was given once daily
  Interventions: Drug: amlodipine plus atorvastatin (Caduet)
- Amlodipine (Norvasc) (Active Comparator): amlodipine(Norvasc, Pfizer, USA) given once daily
  Interventions: Drug: amlodipine (Norvasc)

INTERVENTIONS:
Drug: amlodipine plus atorvastatin (Caduet)
  Arms: Amlodipine Plus Atorvastatin (Caduet)
Drug: amlodipine (Norvasc)
  Arms: Amlodipine (Norvasc)

SUMMARY:
The primary objective of this study is to test the hypothesis that amlodipine plus atorvastatin given in a single tablet (Caduet), compared with amlodipine alone (Norvasc), has a stronger effect in protection of arterial structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men, aged from 40 to 75 years;
2. Women with child-bearing potential should apply an adequate non-pharmacological contraceptive technique;
3. Untreated patients or those on a single antihypertensive drug (except calcium channel blocker ) but with an uncontrolled blood pressure on conventional measurement, ranging from 140 to 179 mm Hg systolic or from 90 to 109 mm Hg diastolic. The conventional blood pressure is the average of 3 consecutive measurements in the sitting position or a single visit.
4. The 24 h ambulatory blood pressure should be at least 130 mm Hg systolic or 80 mm Hg diastolic, or higher;
5. Fasting total cholesterol concentration ranging from 4.14 to 6.22 mmol/L (160 to 240 mg/dL);
6. Endothelium-dependent flow-mediated dilatation (FMD) below 10%;
7. Serum activity of aspartate aminotransferase (AST), alanine aminotransferase (ALT), and creatine kinase (CK) should be within the normal range;
8. Patients should not be on treatment with statins or other lipid-lowering drugs within 3 months of randomization;
9. The patients should sign the informed consent form prior to the participation in the trial at the first visit;
10. Patients should be independent and likely to adhere to the study protocol.

Exclusion Criteria:

1. Secondary hypertension;
2. Low-density lipoprotein cholesterol (LDL-C) below 2.59 mmol/L (100mg/dL);
3. Renal dysfunction defined as eGFR<60ml/min/1.73m2;
4. Current treatment with specific drugs or diets, such as fibrates (especially gemfibrozil), verapamil, amiodarone, grapefruit juice;
5. Excessive alcohol consumption defined as drinking more than 1L/day;
6. Stroke within 2 years of randomization or myocardial infarction occurred previous;
7. Known contra-indications to a dihydropyridine calcium channel blocker or statins;
8. Any life threatening condition;
9. Current participation in another trial or trials.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
flow-mediated dilation (FMD) | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.

SECONDARY OUTCOMES:
pulse wave velocity (cf-PWV, ba-PWV) | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.
liver function | 6-24weeks
  After 6-week maintenance treatment or at 24-week final visit.
  Intolerable adverse events which may or may not be related to the trial treatment, including:
  1. Levels of AST or ALT more than three times the upper limit of normal;
  2. Myalgia symptoms appear with no or only a moderate increase in CK (3 to 10 times above upper limit of normal), but repeated measurements of CK is progressively increasing;
  3. Myalgia symptoms appear, the concentration of CK is 10 times higher than the upper limit of normal.
ankle-brachial index (ABI) | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.
augmentation index (AIx) | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.
carotid intima-media thickness (IMT) | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.
cholesterol level | 12-24 weeks
  After 12-week maintenance treatment or at 24-week final visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Hypertension, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Pingjin Gao